CLINICAL TRIAL: NCT01312636
Title: A Multicentre, Open Label, Observational, Non-interventional Study to Evaluate Safety and Efficacy of NovoSeven® in Patients With Congenital FVII Deficiency - Registry for All Treated Patients
Brief Title: Observational Study on Safety and Efficacy of NovoSeven® in Subjects With Congenital FVII Deficiency
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: F7HAEM-3862; U1111-1116-1529 (Other: WHO)
Record Dates: First submitted 2011-03-02; First posted 2011-03-11 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Congenital Bleeding Disorder; Congenital FVII Deficiency

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: activated recombinant human factor VII

INTERVENTIONS:
Drug: activated recombinant human factor VII — Data will be collected at the baseline visit and approximately once a year until end of study.

SUMMARY:
This study is conducted in Japan. The aim of this observational study is to evaluate the long-term safety and efficacy of activated recombinant human factor VII (NovoSeven®) in subjects with congenital FVII deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Congenital FVII deficiency
* Never been treated with NovoSeven® before
* Patients already in treatment with NovoSeven®

Exclusion Criteria:

* History of hypersensitivity to any of the components in NovoSeven®

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All subjects with a FVII deficiency to whom activated recombinant human factor VII (NovoSeven®) is administered
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2011-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Presence and/or the appearance of inhibiting antibodies to factor VII and/or therapy-related thrombosis on using NovoSeven® under normal clinical practice conditions | once a year in years 1-4

SECONDARY OUTCOMES:
To assess the treatment evaluation for bleeding episodes | year 1, year 4
To assess the course and outcome of pregnancy in women treated with novoseven | until 1 month after giving birth

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Tokyo, Japan

REFERENCES:
- [Derived] Seita I, Kinai E. A multicenter, observational study to evaluate hemostasis following recombinant activated FVII treatment in patients in Japan with congenital factor VII deficiency. Blood Coagul Fibrinolysis. 2023 Jul 1;34(5):295-304. doi: 10.1097/MBC.0000000000001225. Epub 2023 Jun 23. PMID 37395185
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com